CLINICAL TRIAL: NCT04683627
Title: A 12-Week, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase 3 Study to Evaluate the Efficacy and Safety of HP-5000 Topical System (Patch) in Subjects With Osteoarthritis Pain of the Knee
Brief Title: A 12-week Study to Evaluate the Efficacy and Safety of HP-5000 in Subjects With Osteoarthritis Pain of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Noven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Noven Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-5000-US-07
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis Pain of the Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HP-5000 Treatment (Experimental): HP-5000 Topical Patch will be evaluated against placebo topical patches.
  Interventions: Drug: Diclofenac sodium active topical patch
- Placebo Treatment (Placebo Comparator): Placebo patches without diclofenac sodium will be used.
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Diclofenac sodium active topical patch — A topical patch with diclofenac sodium as active ingredient was used and evaluated for the treatment of OA pain of the knee.
  Other Names: HP-5000
  Arms: HP-5000 Treatment
Drug: Placebo patch — A placebo patch without diclofenac sodium was used for the placebo arm.
  Other Names: Placebo
  Arms: Placebo Treatment

SUMMARY:
A 12-week, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase 3 study to Evaluate the Efficacy and Safety of HP-5000 in Subjects with Osteoarthritis (OA) Pain of the Knee

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, and placebo-controlled phase 3 study evaluating the safety and efficacy of HP-5000 in subjects with OA pain of the knees. The study will consist of up to a 28-day Screening Phase that will include a Washout Period of current prescription and over the counter (OTC) analgesics; a 12-week Double-blind Treatment Phase, and a 1-week safety Follow-up Phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 40 to 85 years with a clinical diagnosis of OA of the target knee according to the American College of Rheumatology criteria.
* Has an X-ray of the target knee, taken no more than 1 year before Baseline, showing evidence of OA.
* Has pain of OA in the designated/target study knee.

Exclusion Criteria:

* Body mass index (BMI) > 40.
* Any subject who did not follow the restriction of prohibited therapies during Washout period.
* Arthritis of the target knee that is not caused by OA but caused by diseases such as rheumatoid arthritis, gout, psoriasis, syphilitic arthropathy, ochronosis, metabolic or other primary bone disease, or acute traumatic injury.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Noven Pharmaceuticals, Inc.
Locations (10):
- United States (10):
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Clinical Research of West Florida,Inc., Clearwater, Florida
  - Universal Axon Clinical Research, LLC, Doral, Florida
  - The Arthritis and Diabetes Clinic, Inc., Monroe, Louisiana
  - Noven Pharmaceuticals, Inc., Jersey City, New Jersey
  - Velocity Clinical Research, Cincinnati, Ohio
  - Partners in Clinical Research, Cumberland, Rhode Island
  - Palmetto Clinical Research, Summerville, South Carolina
  - Metroplex Clinical Research Center, Dallas, Texas
  - Quality Research Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant contributed one study knee in this study.
Groups:
- HP-5000 Treatment: Diclofenac Sodium Active Topical Patch was evaluated against the placebo patch for 12-week for the treatment of OA pain of the knee
- Placebo Treatment: Placebo topical patch
Period: Overall Study
Arm/Group | HP-5000 Treatment | Placebo Treatment
Started | 184 | 186
Completed | 184 | 185
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HP-5000 Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 184 | 185 | 369
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 111 | 120 | 231
  >=65 years | 73 | 65 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (8.62) | 61.4 (8.94) | 61.8 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 122 | 241
  Male | 65 | 63 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 57 | 115
  Not Hispanic or Latino | 124 | 128 | 252
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 29 | 22 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 27 | 57
  White | 124 | 135 | 259
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 184 | 185 | 369
Duration of OA of the knee [Mean (Standard Deviation); unit: years] | 7.4 (6.42) | 8.7 (8.81) | 8.0 (7.73)
BMI [Mean (Standard Deviation); unit: Kg/m2] | 30.49 (5.004) | 30.06 (5.166) | 30.28 (5.083)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in WOMAC Pain Score (Intent-to-treat Set)
Description: To evaluate efficacy of HP-5000 patch treatment compared with HP-5000 placebo patch treatment of Osteoarthritis of the knee as evaluated by change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score from baseline to week 12. WOMAC pain score is a scale that evaluate five items including walking, stair climbing, nocturnal, rest and weight bearing. Each item is rated on a scale of 0 to 4, with 0 being no difficulty and 4 being extremely difficulty. The total score is the sum of five items. The total score ranges from 0 to 20 with a low score considered a better outcome and a high score considered a worse outcome.
Time Frame: Baseline and 12-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HP-5000 Treatment | Placebo Treatment
Number analyzed (Participants) | 184 | 185
score on a scale | -4.6 (0.26) | -5.4 (0.26)

2. Secondary Outcome: Change From Baseline to Week 12 in WOMAC Stiffness Score
Description: as for outcome 1
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo Treatment: Placebo topical patch was applied to the target knee on subjects with Osteoarthritis of the knee(s) for 12-week treatment.
Arm/Group | HP-5000 Treatment | Placebo Treatment
Number analyzed (Participants) | 184 | 185
score on a scale | -1.6 (0.12) | -1.8 (0.12)

3. Secondary Outcome: WOMAC Physical Function Change From Baseline at Week 12
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HP-5000 Treatment | Placebo Treatment
Number analyzed (Participants) | 184 | 185
score on a scale | -13.3 (0.80) | -15.9 (0.89)

ADVERSE EVENTS:
Time Frame: up to 13 weeks
Description: The safety population includes all subjects who have at least 1 patch of double-blind study drug applied and who have a at least 1 post-dose safety measurement during the double-blind treatment phase.
Arm/Group | HP-5000 Treatment | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/184 | 4/185
Serious Adverse Events (participants affected / at risk) | 0/184 | 4/185
Other Adverse Events (participants affected / at risk) | 33/184 | 46/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HP-5000 Treatment (N=184) | Placebo Treatment (N=185)
Atrial Fibrillation (Cardiac disorders) | 0 | 1
vertigo (Ear and labyrinth disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HP-5000 Treatment (N=184) | Placebo Treatment (N=185)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Sinus bradycardia (Cardiac disorders) | 3 | 2
Atrioventricular block first degree (Cardiac disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 3
Application site dryness (General disorders) | 1 | 2
application site rash (General disorders) | 0 | 3
Application site swelling (General disorders) | 1 | 2
Application site vesicles (General disorders) | 3 | 0
Pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 1
Application site Bruise (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
Covid-19 (Infections and infestations) | 4 | 3
Urinary tract Infection (Infections and infestations) | 3 | 3
Sinusitis (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2
Hepatic enzyme increased (Investigations) | 2 | 1
Hpokalaemia (Metabolism and nutrition disorders) | 0 | 2
osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT04683627/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT04683627/SAP_003.pdf